CLINICAL TRIAL: NCT00632697
Title: Combined Laparoscopic Surgery and Pentoxifylline Therapy for Treatment of Endometriosis-Associated Infertility: A Preliminary Study
Brief Title: Pentoxifylline and Endometriosis
Acronym: LETS1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LETS
Record Dates: First submitted 2008-03-04; First posted 2008-03-11 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Endometriosis-Associated Infertility
Keywords: endometriosis; immunomodulation; infertility; laparoscopic surgery; pentoxifylline
MeSH Terms: conditions — Endometriosis; Infertility | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: pentoxifylline
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pentoxifylline — 800 mg daily for six months
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
To prove efficacy of an immunomodulator called pentoxifylline in the treatment of endometriosis in infertile patients undergoing laparoscopy surgery

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients having early endometriosis as the only factor of their infertility

Exclusion Criteria:

* Previous treatment for endometriosis or patients having pelvic disorders in addition to endometriosis

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2001-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 6 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Creus M, Fabregues F, Carmona F, del Pino M, Manau D, Balasch J. Combined laparoscopic surgery and pentoxifylline therapy for treatment of endometriosis-associated infertility: a preliminary trial. Hum Reprod. 2008 Aug;23(8):1910-6. doi: 10.1093/humrep/den167. Epub 2008 May 16. PMID 18487215